CLINICAL TRIAL: NCT03103750
Title: Vitamin D as a Therapeutic Adjunct in the Stimulant Treatment of ADHD: a Proof-of-concept Study of Stimulant-induced Dopamine Release Using [11C]-PHNO PET in Healthy Humans
Brief Title: Vitamin D as a Therapeutic Adjunct in the Stimulant Treatment of ADHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Brain & Behavior Research Foundation (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000020604; M# 25288 (Other Grant/Funding Number: Brain and Behavior Research Foundation); 1R01AT010508-01A1 (NIH)
Record Dates: First submitted 2017-03-30; First posted 2017-04-06 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: ADHD
Keywords: Vitamin D
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Magnetic Resonance Spectroscopy; Calcitriol; Dextroamphetamine

STUDY DESIGN:
Intervention Model Description: This is a within-subject, two-day four-scan, randomized, double-blind, placebo-controlled study design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Calcitriol then placebo (Experimental): Healthy volunteers will receive a baseline MRI. On the night before and day of testing, subjects will receive two doses of calcitriol (3.0mcg total), followed by PHNO injection and PET Scan #1. After PET Scan #1, subjects will receive a Dexedrine dose, followed by PHNO injection and PET Scan #2. A minimum of six days later, subjects will receive two doses of placebo for the night before and day of testing, followed by a third PHNO injection and PET scan #3. After PET scan #3, subjects will receive another Dexedrine dose, followed by PHNO injection and PET scan #4.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Drug: PHNO; Dietary Supplement: calcitriol; Drug: Placebo oral capsule; Procedure: high-resolution research tomography; Drug: Dextro Amphetamine
- Placebo then Calcitriol (Experimental): Healthy volunteers will receive a baseline MRI. On the night before and day of testing, subjects will receive two doses of placebo, followed by PHNO injection and PET Scan #1. After PET Scan #1, subjects will receive a Dexedrine dose, followed by PHNO injection and PET Scan #2. A minimum of six days later, subjects will receive two doses of calcitriol (3.0mcg total) for the night before and day of testing, followed by a third PHNO injection and PET scan #3. After PET scan #3, subjects will receive another Dexedrine dose, followed by PHNO injection and PET scan #4.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Drug: PHNO; Dietary Supplement: calcitriol; Drug: Placebo oral capsule; Procedure: high-resolution research tomography; Drug: Dextro Amphetamine

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Magnetic resonance imaging (MRI) scans (3 T) will be collected in each subject for the purposes of excluding participants with anatomical abnormalities and anatomically co-registering PET and MRI for image analysis
Drug: PHNO — Used as a tracer for in vivo imaging.
Dietary Supplement: calcitriol — three 0.5 mcg capsules
Drug: Placebo oral capsule — three 0.5 mcg capsules
Procedure: high-resolution research tomography — A functional imaging technique that is used to observe metabolic processes in the body.
  Other Names: PET scan
Drug: Dextro Amphetamine — Dexedrine 0.3 mg/kg, to a maximum dose of 30 mg
  Other Names: Dexedrine

SUMMARY:
Specific Aim 1: As part of a within-subject, two-days, study design, to determine whether acute calcitriol (vs. placebo) pre-treatment is associated with greater amphetamine (Amp)-induced dopamine (DA) release in the caudate, putamen, ventral striatum (VST), and substantia nigra / ventral tegmental area (SN/VTA) of healthy human subjects.

Specific Aim 2: To determine whether acute calcitriol (vs. placebo) pre-treatment is associated with better performance on a test of attention (e.g., the Continuous Performance Task or CPT-IP), after treatment with amphetamine. Hypothesis: Investigators hypothesize that Subjects pre-treated with calcitriol will have faster reaction times/higher accuracy on the CPT-IP vs. subjects pre-treated with placebo, after treatment with amphetamine.

DETAILED DESCRIPTION:
Increases in the rates of childhood ADHD over the past two decades have lead to speculation that calcitriol deficiency (e.g., secondary to the increased use of sunscreen and/or increases in sedentary, indoor lifestyles in children) plays a causal/contributory role in the etiology of ADHD. To date, evidence of a direct link is lacking. One study showed higher maternal circulating Vitamin D levels in pregnancy are associated with lower risk of developing ADHD-like symptoms in childhood. On the other hand, another study did not replicate the above association, and a prospective study using umbilical cord samples stored at the time of birth reported no difference in serum vitamin D levels between ADHD group versus healthy controls. In terms of clinical trials, one randomized double blind study among adults with ADHD reported a beneficial effect of the intervention, measured with the Conners Adult ADHR rating scale, in comparison with placebo, but the intervention included the combination of vitamin D and several other micronutrients. An analysis of moderators of a positive response to ADHD behaviors did not reveal a significant predictive effect of vitamin D.

However, recent studies provide intriguing indirect evidence of an inverse relationship between solar intensity (SI) and/or altitude (a proxy for greater sun/UV light exposure) and regional rates of ADHD. One study examined three large datasets across 49 U.S. states for 2003 and 2007, and across 9 non-U.S. countries. This study examined the prevalence of ADHD and Solar Intensity (SI) maps. They found an inverse association between solar intensity and prevalence of ADHD. Another study examined two national survey datasets. They found an inverse relationship between altitude and prevalence of ADHD. Investigators hypothesize, as suggested by Huber, that a common denominator on the above studies is the increased vitamin D levels in those exposed to a higher solar intensity, which is known to increase with altitude.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Voluntary, written, informed consent
* Physically healthy by medical history, physical, neurological, ECG, and laboratory examinations
* For females, non-lactating, with a negative serum or urine pregnancy test
* Lab results without clinically relevant findings (e.g. renal function, electrolytes, and vitamin D levels)
* English speaking

Exclusion Criteria:

* Medical contraindication to Dexedrine administration (e.g., history of cardiac problems, seizures, glaucoma, hypertension, hyperthyroidism, etc.)
* Medical contraindication to calcitriol administration (e.g., history of hypersensitivity to calcitriol or any component of the formulation, hypercalcemia or vitamin D toxicity)
* History of substance dependence (e.g., alcohol, opiates, sedative hypnotics), except for nicotine
* A primary major DSM-5 psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) as determined by the Structured Clinical Interview for DSM-5 (SCID)
* A history of significant medical (e.g., cardiovascular, diabetic/metabolic) or neurological (e.g., cerebrovascular accidents, seizure, traumatic brain injury) illness
* Positive answers on the cardiac history questionnaire that may place the subject at higher risk, as determined by an internal medicine specialist or cardiologist's review of both the questionnaire responses and screening ECG
* Current use of psychotropic and/or potentially psychoactive prescription medications
* For females, laboratory (β-HCG) or physical evidence of pregnancy/lactation 9) MRI-incompatible implants and other contraindications for MRI (i.e., aneurysm clip, metal fragments, internal electrical devices such as a cochlear implant, spinal cord stimulator or pacemaker)
* History of claustrophobia or feeling of inability to lie still on his/her back for the PET or MRI scans
* History of any bleeding disorder or current anticoagulant therapy
* Donation or loss of 550 mL of blood or more (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to the first test day.
* Use of any prescription medications and/or over-the-counter medications, vitamins and/or herbal supplements which could have a negative clinical interaction with calcitriol/Dexedrine or which could confound scientific results of the study, within 2 weeks prior to each test day (e.g., thiazide diuretics, Mg based antiacids, digoxin, etc,.).
* Serum levels of 25(OH)D3 below 20 ng/ml.
* Obesity i.e. BMI over 30 (more prone to lower vitamin D levels)
* Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over Radioactive Drug Research Committee (RDRC) limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
* Subjects with current, past or anticipated exposure to radiation in the work place
* History of kidney stones within the past 5 years
* Any degree of renal failure
* History of parathyroid disorder (hyper or hypoparathyroidism)
* History of osteoporosis or any pathologic fractures
* Vitamin D supplementation in any form in the past 3 months
* Known hypersensitivity to Dexedrine, [11C]PHNO, or calcitriol
* Malabsorption syndromes (i.e. Celiac sprue)
* Serum corrected calcium > 10.5 mg/dl or phosphate > 4.2 mg/dl

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, PhD, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcitriol Then Placebo | Placebo Then Calcitriol
Started | 12 | 12
Completed First Leg of Crossover | 8 | 10
Completed | 8 | 10
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — PET Equipment Related | 2 | 2

BASELINE CHARACTERISTICS:
Population: Overall sample prior to randomization to crossover sequence.
Groups:
- Overall Participants: Baseline characteristics of all participants prior to group order randomization.
Arm/Group | Overall Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.96 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Non-displaceable Tracer Binding Potentials
Description: non-displaceable tracer binding potentials (BPND = VT - VREF / VREF), which are linearly proportional to the density of available D2/3 Rs, computed using a simplified reference tissue model (SRTM) utilizing the cerebellum as a reference region.
Time Frame: day 1
Population: Participants required complete imaging data (i.e., 4/4 completed PET scans and a completed MRI) in order to be included in analysis. Thus, only n = 18 participants were analyzed to assess BPND.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Calcitriol: Healthy volunteers will receive a baseline MRI. On the night before and day of testing, subjects will receive two doses of calcitriol (3.0mcg total), followed by PHNO injection and PET Scan #1. After PET Scan #1, subjects will receive a Dexedrine dose, followed by PHNO injection and PET Scan #2. A minimum of six days later, subjects will receive two doses of placebo for the night before and day of testing, followed by a third PHNO injection and PET scan #3. After PET scan #3, subjects will receive another Dexedrine dose, followed by PHNO injection and PET scan #4.
  Magnetic Resonance Imaging (MRI): Magnetic resonance imaging (MRI) scans (3 T) will be collected in each subject for the purposes of excluding participants with anatomical abnormalities and anatomically co-registering PET and MRI for image analysis
  PHNO: Used as a tracer for in vivo imaging.
  calcitriol: three 0.5 mcg capsules
  high-resolution research tomography: A functional imaging technique that is used to observe metabolic processes in the body.
  Dextro Amphetamine: Dexedrine 0.3 mg/kg, to a maximum dose of 30 mg
- Placebo: Healthy volunteers will receive a baseline MRI. On the night before and day of testing, subjects will receive two doses of placebo, followed by PHNO injection and PET Scan #1. After PET Scan #1, subjects will receive a Dexedrine dose, followed by PHNO injection and PET Scan #2. A minimum of six days later, subjects will receive two doses of calcitriol (3.0mcg total) for the night before and day of testing, followed by a third PHNO injection and PET scan #3. After PET scan #3, subjects will receive another Dexedrine dose, followed by PHNO injection and PET scan #4.
  Magnetic Resonance Imaging (MRI): Magnetic resonance imaging (MRI) scans (3 T) will be collected in each subject for the purposes of excluding participants with anatomical abnormalities and anatomically co-registering PET and MRI for image analysis
  PHNO: Used as a tracer for in vivo imaging.
  Placebo oral capsule: three 0.5 mcg capsules
  high-resolution research tomography: A functional imaging technique that is used to observe metabolic processes in the body.
  Dextro Amphetamine: Dexedrine 0.3 mg/kg, to a maximum dose of 30 mg
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 8 | 10
ratio
  Region of interest: Ventral Striatum | 2.93 (0.63) | 2.91 (0.32)
  Region of interest: Caudate | 1.50 (0.30) | 1.50 (0.19)
  Region of interest: Putamen | 2.21 (0.47) | 2.21 (0.26)
  Region of interest: Substantia Nigra/Ventral Tegmental Area | 0.92 (0.30) | 1.01 (0.24)

2. Primary Outcome: Non-displaceable Tracer Binding Potentials
Description: as for outcome 1
Time Frame: day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 10 | 8
ratio
  Region of interest: Ventral Striatum | 2.91 (0.32) | 3.05 (0.66)
  Region of interest: Caudate | 1.52 (0.21) | 1.59 (0.30)
  Region of interest: Putamen | 2.31 (0.28) | 2.38 (0.47)
  Region of interest: Substantia Nigra/Ventral Tegmental Area | 1.08 (0.25) | 1.07 (0.31)
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; The primary hypothesis of calcitriol-related differences in amphetamine-induced dopamine release was determined by significance of the main effect of medication (calcitriol vs. placebo) on %change in BPND (i.e., post-Amp relative to pre-Amp scans) at a threshold of p<0.05; Test type: Superiority; p = 0.016, Mixed Models Analysis

3. Secondary Outcome: Continuous Performance Task (CPT-IP)
Description: In this computer based test, subjects are shown a random sequence of numbers (2-digit, 3-digit, and 4-digit) and are instructed to press a button as quickly and accurately as possible (with their preferred hand) when a number repeats. Subjects are instructed to withhold their response for any other sequence of numbers. The measure is presented as dprime, which is calculated: d' = z(H) - z(F), where z(H) is the z-score of the hit rate and z(F) is the z-score of the false positive rate. A z-score of 0 represents the population mean. d' is indicates better performance on the task with higher values, z(H) indicates better performance on the task with higher values due to higher hit rate, and z(F) indicates worse performance on the task with higher values due to higher false positive rates.
Time Frame: day 1
Population: All participants completed both study arms
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 8 | 10
z-score | 3.03 (0.74) | 3.35 (1.22)

4. Secondary Outcome: Continuous Performance Task (CPT-IP)
Description: as for outcome 3
Time Frame: day 7
Population: All participants completed both study arms.
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 10 | 8
z score | 3.03 (0.74) | 3.22 (0.42)
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; Test type: Superiority; p = 0.55, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: Adverse events were collected at the individual level and were not distinguished at the stage of the crossover.
Arm/Group | Calcitriol Then Placebo | Placebo Then Calcitriol
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcitriol Then Placebo (N=12) | Placebo Then Calcitriol (N=12)
Mild transient nausea (Gastrointestinal disorders) | 4 | 4
Mild anxiety (Psychiatric disorders) | 1 | 0
Mild insomnia (General disorders) | 2 | 2
Nausea and vomiting (Gastrointestinal disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Asymptomatic non-exclusionary bradycardia (Cardiac disorders) | 0 | 1
Hypertension, asymptomatic and non-exclusionary (Vascular disorders) | 1 | 0
Throat irritation (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03103750/Prot_SAP_000.pdf